CLINICAL TRIAL: NCT03744013
Title: A Post Market Prospective Study of FORTIVA® 1mm Porcine Dermis in Breast Reconstruction
Brief Title: A Post Market Prospective Study of FORTIVA® 1mm Porcine Dermis
Acronym: APPeaR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1104
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Mammoplasty

STUDY DESIGN:
Intervention Model Description: post market prospective, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perforated (Active Comparator): Fortiva® 1mm perforated ADM
  Interventions: Device: Fortiva® 1mm
- Non-perforated (Active Comparator): Fortiva® 1mm non-perforated ADM
  Interventions: Device: Fortiva® 1mm

INTERVENTIONS:
Device: Fortiva® 1mm — Post mastectomy immediate reconstruction

SUMMARY:
This is a post market prospective, multi-center study of up to 100 subjects undergoing post-mastectomy breast reconstruction (50 Fortiva® 1mm perforated and 50 Fortiva® 1mm non-perforated) at up to 10 clinical study sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Female 18 years or older
2. A candidate for immediate breast reconstruction during post-skin sparing or nipple-sparing mastectomy (unilateral or bilateral)
3. Estimated life expectancy > 2 years
4. Able and willing to return for all scheduled and required study visits
5. Able to provide written informed consent for study participation
6. Able to read, understand and complete study questionnaires

Exclusion Criteria:

1. Any of the conditions listed in the approved labeling as contraindicated
2. Currently enrolled or plans to enroll in another clinical study that would affect the validity of the study
3. Any patient that per the physician's judgement is not a good candidate for this study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Safety of Fortiva® tissue matrix | 24 months
  Safety will be evaluated by assessing the incidence of device and/or procedure related adverse events.
Performance of Fortiva® tissue matrix | 24 months
  • Analysis of the subject's overall satisfaction with the breast reconstruction procedure will be assessed by obtaining subject's perception of the outcomes using the Breast-QTM - Reconstruction survey.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (4):
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Frankfurt University Hospital, Frankfurt am Main
  - University Hospital Technical University, Munich, München
  - University Hospital, Ulm, Ulm
- United Kingdom (2):
  - Guy's Hospital, London
  - Nightingale Breast Unit, Manchester University NHS Foundation Trust (MFT), Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No